CLINICAL TRIAL: NCT01373840
Title: Role of Dopamine Receptors in Primary Focal Dystonias
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 201102481
Record Dates: First submitted 2011-06-10; First posted 2011-06-15 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Healthy; Focal Dystonias
Keywords: focal; dystonia; dopamine; receptor
MeSH Terms: conditions — Dystonic Disorders; Dystonia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- healthy controls
- patients with focal dystonias

SUMMARY:
Dystonia is a disabling movement disorder characterized by repetitive patterned or sustained muscle contractions causing twisting or abnormal postures that may afflict 250,000 people in the U.S. While the pathophysiology of dystonia remains uncertain the treatment is rather rudimentary. A better understanding of neural mechanisms of dystonias is not only an invaluable prerequisite for developing better treatment options but also a step toward better understanding of the complex network of basal ganglia. In this study I will investigate if there is any difference between the dopamine receptors and dopamine in people with dystonia and healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age >20
* Male or Female
* Any race or ethnicity
* Primary focal dystonia (arm or cranial)
* Ability to give informed consent

Exclusion criteria:

* Family history of dystonia
* Pregnancy (confirmed with negative urine pregnancy test in women of child bearing potential), breastfeeding
* Exposure to radiation therapy
* Any MRI contraindications such as foreign metallic implants, pacemaker, and aneurysm clip etc.
* History of cardiac disease, uncontrolled hypertension, abnormal EKG during screening phase
* History of exposure to any drugs affecting dopaminergic systems within the last 6 months (e.g. dopamine receptor blocking agents, cocaine, amphetamine, tetrabenazine, reserpine, L-dopa, dopamine agonists, as they might affect the dopamine receptor binding or endogenous dopamine).
* Active depression (Beck Depression Inventory_II >14)
* Cognitive impairment (Mini-Mental State Score <27)
* CNS active medications such as gabapentin or narcotics, muscle relaxants which might be given for pain in the 3 days prior to study
* History of stroke, seizure, cerebral palsy, generalized dystonia, parkinsonism, inability to hold head still during the scanning time.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any healthy control or patient with primary focal dystonia or arm or face.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2011-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Perlmutter Joel, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States